CLINICAL TRIAL: NCT05505500
Title: Preparing a Clinical Outcomes Assessment Set for Nephrotic Syndrome
Brief Title: Interview Study of Adult and Child Patients and Parents of Children With Swelling Due to Nephrotic Syndrome.
Acronym: Prepare-NS
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Northwestern University (Other); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Eloise Salmon, Assistant Professor of Pediatrics, Division of Nephrology, University of Michigan
Other Study IDs: HUM00208148; 5UG3FD007308-02 (FDA)
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Fluid Overload; Glomerulosclerosis, Focal Segmental; Edema; Membranous Nephropathy; Minimal Change Disease; Minimal Change Nephrotic Syndrome; IgM Nephropathy; Nephrotic Syndrome; Glomerular Disease; Nephrotic Syndrome, Minimal Change; Nephrotic Syndrome in Children; Nephrotic Syndrome With Edema (Diagnosis); FSGS
Keywords: Nephrotic Syndrome; Child; Adult; Fluid Overload; Edema; FSGS; Minimal Change Disease; Membranous Nephropathy; IgM Nephropathy
MeSH Terms: conditions — Edema; Glomerulosclerosis, Focal Segmental; Glomerulonephritis, Membranous; Nephrosis, Lipoid; Nephrotic Syndrome; Disease | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parent/Guardian of child with Nephrotic Syndrome (NS): This group will help create the Observer Reported Outcome (ObsRO) tool.
  Interventions: Behavioral: Interview
- Person with Nephrotic Syndrome (NS): This group will help create the Patient Reported Outcome (PRO) tool.
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Concept Elicitation Interviews are used to create tools followed by Cognitive Debrief Interviews that are used to review created tools.

SUMMARY:
Researchers from the University of Michigan and Northwestern University are studying people's experiences with swelling caused by Nephrotic Syndrome. Interviews with patients (child and adult) and parents of young children will be conducted. The information collected from the interviews will be used to develop a survey to use when testing new medications for Nephrotic Syndrome.

Please consider participating in a 1-hour long interview with the Prepare-NS research study to discuss children and adults experiences with swelling.

DETAILED DESCRIPTION:
This registration includes concept elicitation, analysis and creation of complementary survey measures focused on edema/fluid overload of nephrotic syndrome. The measures to be developed include an Observer Reported Outcome (ObsRO) and Patient Reported Outcome (PRO). The ObsRO and PRO substudies are Institutional Review Board (IRB) approved at release.

The researcher's goal is to produce core outcome sets of patient-rated and observer reported Fluid Overload (edema) measures that can be applied across the fluid overload severity continuum, fit to help drug development in this area.

ELIGIBILITY:
Criteria for the Observer Reported Outcomes (ObsRO) cohort of the study:

Inclusion Criteria:

1. Parents/guardians must be able to read and understand English;
2. Parents/guardians must be caring for a child (ages 2-11.999) with a medically documented diagnosis of idiopathic (primary) Nephrotic Syndrome (NS) or primary or monogenic NS associated kidney disease. Populations with Primary NS Conditions: Focal segmental glomerulosclerosis (FSGS), Minimal Change Disease (MCD), Immunoglobulin M (IgM) Nephropathy, Membranous Nephropathy (MN), and childhood - onset nephrotic syndrome not biopsied;
3. The child must have a current NS-associated edema
4. The child must have native kidney function
5. Parents/guardians must provide informed consent.

Exclusion Criteria:

1. Index case with dialysis dependence throughout the 3-month pre-enrollment period

Criteria for the Patient Reported Outcomes (PRO) cohort of the study:

Inclusion Criteria:

1. ≥8 years of age
2. Able to read and understand English
3. Primary (idiopathic) kidney disease that causes NS or monogenic NS associated kidney disease.

   i. Populations with Primary Nephrotic Syndrome (NS) Conditions include: FSGS, MCD, IgM nephropathy, MN, and childhood - onset nephrotic syndrome not biopsied
4. Current NS-associated edema
5. Kidney function with most recent estimated Glomerular Filtration Rate (eGFR) > 25 ml/min/1.73m2
6. Informed Consent: For patients ≥8 to <18 years of age: a parent or legal guardian provide informed consent and the patient must provide assent. Patients ≥18 years of age must provide informed consent.

Exclusion Criteria:

1. Native kidney disease participant with dialysis dependence during the 3-month pre-enrollment period
2. Co-existing significant chronic or severe acute health condition that has the potential to influence how the participant feels or functions as related to fluid overload in NS

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ObsRO Study Population: Data collection will involve approximately 20-40 parents/guardians of children ages 2-11.999 with NS
  PRO Study Population: Data collection will involve N = 60 to 95 patients ≥8 years of age with NS (depending on when concept saturation is achieved; see section 9.0 Statistical Considerations for more detail). Recruitment of patients with NS will occur across the United States. Enrollment will take place at the University of Michigan.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Impact of Fluid Overload on symptoms and functioning | Interviews are 60 minutes
  Themes generated through qualitative analysis from semi-structured interviews
Observer Reported Impact of Fluid Overload on symptoms and functioning | Interviews are 60 minutes
  Themes generated through qualitative analysis from semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Eloise Salmon, M.D., Principal Investigator — University of Michigan; John Peipert, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No